CLINICAL TRIAL: NCT05164822
Title: Evolution of Neuropathies Associated With Necrotizing Vasculitis: Prospective, Non-interventional, Multicentric Study
Brief Title: Evolution of Neuropathies Associated With Necrotizing Vasculitis
Acronym: NERF-VASC
Status: Terminated | Type: Observational
Why Stopped: insufficient number of inclusions
Sponsor: Lille Catholic University (Other)
Collaborators: UNEOS (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC-P0092
Record Dates: First submitted 2021-10-21; First posted 2021-12-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Necrotizing Vasculitis; Neuropathy
Keywords: Necrotizing Vasculitis; Neuropathy; Score development; Evolution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Necrotizing Vasculitis: Patient with an initial diagnosis or a relapse of :
  - Systemic Vasculitic Neuropathy (SVN): Primary Necrotizing Vasculitis answering the Chapel Hill Consensus Conference criteria associated with a symptomatic Vasculitic Peripheral Neuropathy
  Or
  - Non Systemic Vasculitic Neuropathy (NSVN): pure symptomatic peripheral neurological impairment without systemic visceral impairment
  Interventions: Other: Necrotizing Vasculitis

INTERVENTIONS:
Other: Necrotizing Vasculitis — Pain scale Diagnosis of necrotizing vasculitis and peripheral neuropathy, Clinical characteristics of the disease, Biological analysis, Treatment and evolution of the disease,
  Questionnaires :
  Neuropathy Impairment Score (NIS) sensitive sub-questionnaire that measures extremity sensitivity.
  MRC (Medical Research Council), which evaluates three motor functions on each member.
  RODS questionnaire on the relationship between your daily activities and your health.
  BVAS (Birmingham Vasculitis Activity Score) disease activity questionnaire. VDI (Vasculitis Damage Index) questionnaire evaluates the sequelae of the disease.
  Rankin Score modified to measure the degree of disability
  Two tests will be performed:
  EMG (electromyogram) to evaluate the electrical activity of the muscles, Walking Test of 10 meters which aims to measure the time taken to travel 10 meters.

SUMMARY:
Necrotizing Vasculitis are inflammatory diseases of the wall of vessels. Neurological damage of the peripheral nerve varies from 7% to 50% of cases depending on the type of Necrotizing Vasculitis.

Peripheral neurological impairment is rarely life threatening (except when associated with other visceral impairment which, in turn, require urgent management with a severity score defined by the Five Factor Score) but impacts the functional outcome by sequelae evaluated by the Vascular Disease Index (VDI).

Four retrospective studies were published with low number of participants, and also mix subgroups of vasculitis Anti-Neutrophil Cytoplasmatic Antibodies (ANCA)+/- GPA (Granulomatosis with polyangiitis), Eosinophilic granulomatosis with polyangiitis (EGPA), Microscopic polyangiitis (MPA), Polyarteritis nodosa (PAN), and Non Systemic Vasculitic Neuropathy (NSVN) and Systemic Vasculitic Neuropathy (SVN).

Overall, management of Necrotizing Vasculitis has evolved significantly over the last two decades, with a dramatic improvement in survival, thanks to new therapeutic strategies and medications. Five-year survival increased from 85% for diagnoses made between 1990 and 1999 to 94.5% for diagnoses made after 2010 Evaluation of relapses of vasculitis, late macro vascular complications, medical-economic evaluation of therapeutic strategies and functional impairment of neuropathies are at the heart of current medical concerns with a view to improve vital and functional prognosis.

Various tests for the evaluation of peripheral neurological damage appear to be relevant tools in vasculitis, although they are not specific: Muscular force scale Medical research council (MRC), Rasch-built overall disability scale (RODS), Inflammatory Neuropathy Cause and Treatment (INCAT) disability score, Construction and validation of the chronic acquired polyneuropathy patient-reported index (CAP-PRI), Health-Related Quality of Life (HR QOL), Medical Interview Satisfaction Scale (MISS), Neuropsychological Impairment Scale (NIS) associated to results of repeated Electromyography.

In this study, MRC, NIS and RODS measurements were chosen for their reproducibility and practicality.

In addition to the immediate or relapse mortality factors assessed by the five-factor score (FFS), a functional morbidity score specific to neuropathies related to necrotizing vasculitis must be developed, as well as the determination of the neurosensory disorders and macro-vascular complications. Therefore it is proposed in this observational study to determine the factors that can be predictive of the functional evolution, in order to build a risk score.

ELIGIBILITY:
Inclusion Criteria:

Adult patient with an initial diagnosis or a relapse of :

- Systemic Vasculitic Neuropathy (SVN): Primary Necrotizing Vasculitis answering the Chapel Hill Consensus Conference criteria associated with a symptomatic Vasculitic Peripheral Neuropathy

Or

- Non Systemic Vasculitic Neuropathy (NSVN): pure symptomatic peripheral neurological impairment without systemic visceral impairment

Exclusion Criteria:

* Symptomatic peripheral neurological impairment not attributable exclusively to primary necrotizing vasculitis
* Diabetes
* Chronic ethylism
* AL (immunoglobulin light chain) amyloidosis or TTR (transthyretin)
* Genetic neuropathies
* Toxic neuropathies
* Sequelae of sciatica
* Opposition to participation in the study
* Lack of social security
* Under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with an initial diagnosis or a relapse of :
  - Systemic Vasculitic Neuropathy (SVN): Primary Necrotizing Vasculitis answering the Chapel Hill Consensus Conference criteria associated with a symptomatic Vasculitic Peripheral Neuropathy
  Or
  - Non Systemic Vasculitic Neuropathy (NSVN): pure symptomatic peripheral neurological impairment without systemic visceral impairment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Time to remission | 24 months
  The time to remission will be collected. Remission is defined by the absence of new symptoms or lesions due to persistent vasculitis activity and the absence of an inflammatory syndrome
Medical Research Council (MRC) score | 24 months
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
  The patient's effort is graded on a scale of 0-5:
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed.
Neuropathy impairment score (NIS) | 24 months
  This score will measure the ankle reflex 0 = normal,
  1. = present with reinforcement,
  2. = absent
Rasch-built Overall Disability (R-ODS) Scale | 24 months
  The R-ODS is a linearly weighted scale developed to capture activity and social participation limitations. Score is between 0 and 48 being 0 the worst and 48 the best one.

SECONDARY OUTCOMES:
Correlation coefficient between gravity factors, impact on daily life and dependence | 24 months
  The Correlation coefficient between severity factors, impact on daily life and dependence will be assessed by a mixed model
Response to treatment | 3, 6, 9, 12 and 24 months
Prevalence of peripheral neurological disorders | 24 months
  Peripheral neurological disorders will be detected by electromyogram
Prevalence of necrotizing vasculitis | 24 months
  Necrotizing vasculitis will be detected by electromyogram
Time to recovery | 24 months
Medical Research Council (MRC) in patients in remission | 24 months
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
  The patient's effort is graded on a scale of 0-5:
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed.
Neuropathy impairment score (NIS) in patients in remission | 24 months
  This score will measure the ankle reflex as follows:
  0 = normal,
  1. = present with reinforcement,
  2. = absent
Rankin score in patients in remission | 24 months
  This scale is used to categorize the level of functional independence. The scale is between 0 and 5 being 0 without symptoms and 5 meaning severe disability.
  0 No symptoms
  1. No significant disability despite symptoms; able to perform all usual tasks and activities.
  2. Mild disability: unable to perform all previous activities, but able to attend to own affairs without assistance.
  3. Moderate disability: requires assistance, but able to walk without assistance.
  4. Moderately severe disability: unable to walk without assistance and unable to care for own bodily needs without assistance.
  5. Severe disability: bedridden, incontinent and requires constant nursing attention and care.
Birmingham Vasculitis Activity Score (BVAS) in patients in remission | 24 months
  BVAS is a validated tool for assessment of disease activity in patients with many different forms of vasculitis (21-23). The BVAS includes scored items grouped into 9 organ systems which capture a broad spectrum of clinical manifestations from vasculitis. Scores can range from 0 to 63 being 0 the best and 63 the worst.
Visual Analogue Scale (VAS) | 24 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: François Maurier, MD, Study Chair — UNEOS
Locations (40):
- France (40):
  - CHU Angers, Angers
  - Hôpital Pellegrin, Bordeaux
  - CH Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Centre Hospitalier Bourg-en-Bresse, Bourg-en-Bresse
  - CHRU Brest, Brest
  - Hôpital Percy, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU DIjon-Bourgogne, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Hôpital Neurologique Pierre Wertheimer - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - Groupe Hospitalier Sud Ile de France, Melun
  - CHR Metz, Metz
  - UNEOS, Metz
  - Groupe Hospitalier du Havre, Montivilliers
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Pasteur, Nice
  - CHU Bicêtre, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpital Cochin, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Perpignan, Perpignan
  - Hôpital Haut-Lévêque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Saint-Malo, St-Malo
  - CHU Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital de Rangueil, Toulouse
  - Hôpital Pierre-Paul Riquet, Toulouse
  - Centre Hospitalier Bretagne-Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No